CLINICAL TRIAL: NCT04783077
Title: Community-Based Communication Approaches for Blood Donation in Ghana
Acronym: C-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Blood Service Ghana (Other); University of Ghana (Other); Syracuse University (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 326045; UG3HL151599 (NIH)
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Blood Donors
Keywords: Blood donation

STUDY DESIGN:
Intervention Model Description: A pilot stratified randomized control trials of WhatsApp compared to control and docudrama (before/after) among first time donors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- FRD Control (Active Comparator)
  Interventions: Behavioral: Control
- VNRBD Control (Active Comparator)
  Interventions: Behavioral: Control
- FRD WhatsApp (Experimental)
  Interventions: Behavioral: WhatsApp
- VNRBD WhatsApp (Experimental)
  Interventions: Behavioral: WhatsApp
- Docudrama (Experimental)
  Interventions: Behavioral: Docudrama

INTERVENTIONS:
Behavioral: WhatsApp — Participants assigned to the WhatsApp group will receive weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.
  Arms: FRD WhatsApp; VNRBD WhatsApp
Behavioral: Control — Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
  Arms: FRD Control; VNRBD Control
Behavioral: Docudrama — Participants will be exposed to a document-drama related to blood donation.
  Arms: Docudrama

SUMMARY:
DESIGN This pilot study utilizes a mixed-methods approach to develop a novel docu- drama communication strategy, design WhatsApp intervention, evaluate the feasibility of a larger pragmatic randomized controlled trial (RCT) of the two communication strategies and assess acceptability of the communication strategies aimed to increase blood donation among first-time blood donors within the catchment areas of the Southern Zonal Blood Centre (SZBC) in Ghana. In sequence, this pilot study and larger RCT are grounded in the PRECEDE-PROCEED implementation science framework. The pilot study has four components: 1) a qualitative component will be used to design a docu-drama, 2) key informant interviews to guide intervention development, 3) a simultaneous randomized pilot trial will evaluate the feasibility of the larger trial design of communication interventions using WhatsApp compared to control, and 4) a final mixed- methods (quantitative survey and focus groups) assessment of participant views of acceptability, effectiveness, feasibility and cultural appropriateness of the two proposed communication interventions.

OBJECTIVES The three objectives of this pilot study are the careful design of a novel docu- drama communication intervention and WhatsApp intervention, evaluation of the feasibility of a larger RCT of communication strategies, and assessment of participant views of the two proposed communication interventions and control among first time blood donors within the catchment areas of the SZBC.

For the purposes of registration for clinicaltrials.gov only the randomized pilot trial communication interventions using WhatsApp compared to control is reported.

The planned sample size for the pilot RCT is n=128 first-time blood donors.

The study population for the pilot RCT is first-time voluntary non-remunerated blood donors (VNRBD) and family/replacement blood donors (FRD) from the SZBC catchment area.

REGIMEN WhatsApp: Participants assigned to the WhatsApp group will receive weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.

Control: Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years-old
* First-time whole blood donor with the SZBC of the NBSG
* Eligible to donate again
* Consent to participate
* Understands one of English, Twi, or Ga
* Have a smart phone
* Have, or be willing to sign up for an active WhatsApp account

Exclusion Criteria:

• History of more than one lifetime whole blood donation (with any blood centre)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Blood Service Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.

RESULTS

PARTICIPANT FLOW:
Groups:
- FRD: Control: Family Replacement Donors (FRD) assigned to Control: Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
- VNRBD: Control: Voluntary Non-Remunerated Blood Donors (VNRBD) assigned to Control: Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
- FRD:WhatsApp: Family Replacement Donors (FRD) assigned to WhatsApp: Participants assigned to the WhatsApp group will receive weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.
- VNRBD: WhatsApp: Voluntary Non-Remunerated Blood Donors (VNRBD) assigned to WhatsApp: Participants assigned to the WhatsApp group will receive weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.
- Docudrama: Participants will be exposed to a docudrama about blood donation.
Period: Overall Study
Arm/Group | FRD: Control | VNRBD: Control | FRD:WhatsApp | VNRBD: WhatsApp | Docudrama
Started | 34 | 33 | 30 | 33 | 14
Completed | 27 | 30 | 28 | 31 | 14
Not Completed | 7 | 3 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomization was into WhatsApp and Control was stratified by donation type (FRD/VNRBD). A separate group of participants will be invited to a single viewing of a filmed docudrama.
Groups:
- FRD: Control: FRD: Control participants received the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
- VNRBD: Control: VNRBD: Control participants received the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
- FRD: WhatsApp: FRD: WhatsApp participants received weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.
- VNRBD: WhatsApp: VNRBD: WhatsApp participants received weekly messages developed by communication specialists aimed to motivate blood donation, be encouraged to discuss their blood donation experiences, and share their own motivations for donating blood in a moderated, closed group over a six-month duration. The moderator will provide guidelines on acceptable use of WhatsApp in the group, including images they can or cannot share. Participants will also receive standard NBSG communications for first-time donors.
- Docudrama: Participants will be exposed to a docudrama related to blood donation.
- Total: Total of all reporting groups
Arm/Group | FRD: Control | VNRBD: Control | FRD: WhatsApp | VNRBD: WhatsApp | Docudrama | Total
Number analyzed (Participants) | 34 | 33 | 30 | 33 | 14 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.62 (6.21) | 23.33 (6.21) | 25.73 (6.70) | 24.33 (5.64) | 24.00 (4.21) | 25.26 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 16 | 8 | 13 | 6 | 47
  Male | 30 | 17 | 22 | 20 | 8 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Akan | 11 | 19 | 14 | 20 | 7 | 71
  Ewe | 6 | 6 | 2 | 5 | 1 | 20
  Dagbani | 3 | 1 | 0 | 1 | 1 | 6
  Ga/Dangbe | 11 | 4 | 8 | 4 | 2 | 29
  Hausa | 1 | 0 | 3 | 0 | 0 | 4
  Other | 2 | 3 | 3 | 3 | 3 | 14
Region of Enrollment [Number; unit: participants]
  Ghana | 34 | 33 | 30 | 33 | 14 | 144
Marital status [Count of Participants; unit: Participants]
  Single | 22 | 32 | 25 | 31 | 14 | 124
  Married | 12 | 1 | 5 | 2 | 0 | 20
Children [Count of Participants; unit: Participants]
  No; children | 23 | 30 | 20 | 29 | 13 | 115
  Yes; children | 11 | 3 | 10 | 4 | 1 | 29
Home Situation [Count of Participants; unit: Participants]
  I live alone | 13 | 7 | 7 | 9 | 4 | 40
  I am a single parent without child/children | 0 | 2 | 1 | 3 | 0 | 6
  I live with only my husband/wife/partner | 4 | 0 | 1 | 0 | 0 | 5
  I live with my husband/wife/partner and children | 8 | 2 | 6 | 2 | 0 | 18
  I live with my parents/relatives/friends | 9 | 21 | 15 | 19 | 10 | 74
  Other | 0 | 1 | 0 | 0 | 0 | 1
Main Method of Transportation [Count of Participants; unit: Participants]
  Private | 1 | 7 | 1 | 8 | 1 | 18
  Public | 30 | 20 | 27 | 17 | 9 | 103
  Other | 3 | 6 | 2 | 8 | 4 | 23
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Primary school | 1 | 0 | 1 | 0 | 0 | 2
  Junior high school | 1 | 5 | 6 | 2 | 1 | 15
  Senior high school | 14 | 13 | 12 | 13 | 4 | 56
  Diploma | 6 | 1 | 2 | 3 | 2 | 14
  Degree | 10 | 12 | 9 | 12 | 7 | 50
  Postgraduate level | 2 | 2 | 0 | 3 | 0 | 7
Employment [Count of Participants; unit: Participants]
  Student | 5 | 18 | 5 | 15 | 9 | 52
  Out of school and/or unemployed | 6 | 3 | 6 | 1 | 0 | 16
  Homemaker/housewife | 1 | 0 | 0 | 0 | 0 | 1
  Informal/part-time employment | 7 | 3 | 3 | 1 | 0 | 14
  Self-employed | 9 | 1 | 8 | 3 | 3 | 24
  Formal employment | 6 | 8 | 8 | 13 | 2 | 37
Income [Count of Participants; unit: Participants]
  No income | 10 | 18 | 9 | 14 | 9 | 60
  Less than GH 500.00 | 2 | 2 | 2 | 1 | 0 | 7
  GH 500.00-1000.00 | 14 | 3 | 5 | 8 | 1 | 31
  GH 1001.00-2000.00 | 3 | 4 | 4 | 1 | 0 | 12
  GH 2001.00-3000.00 | 0 | 2 | 2 | 3 | 2 | 9
  More than GH 3000.00 | 0 | 0 | 0 | 2 | 1 | 3
  Not sure | 1 | 2 | 2 | 1 | 0 | 6
  Prefer not to say | 4 | 2 | 6 | 3 | 1 | 16
Owns item [Number; unit: participants]
  Car | 3 | 4 | 1 | 7 | 1 | 16
  Motorbike | 3 | 1 | 1 | 1 | 2 | 8
  Bicycle | 6 | 5 | 4 | 5 | 2 | 22
  Television | 27 | 26 | 24 | 25 | 11 | 113
  Refrigerator or deep freezer | 25 | 17 | 27 | 20 | 7 | 96
  Radio | 30 | 21 | 28 | 22 | 6 | 107
  Cooking stove | 24 | 17 | 24 | 20 | 9 | 94
Belongs to a Religious Faith [Count of Participants; unit: Participants]
  Christian | 31 | 32 | 26 | 32 | 13 | 134
  Muslim | 3 | 1 | 4 | 1 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Donation Attempt
Description: Blood donation attempt at any time during follow-up. The planned follow-up (i.e., ﬁnal assessment) was at 6-months and 2 weeks from randomization. However, the local protocol IRB approval lapsed between 25 April 2022 and 23 May 2022 during which time participants were unable to receive WhatsApp messaging. In response, the ﬁnal follow-up window was extended by 34 days for all participants, so the participants in the WhatsApp arm would receive all planned messages.
Time Frame: 6 Months and 34 days
Population: The analyses followed a modiﬁed intention-to-treat (mITT) approach. Individuals who consented, were randomized and not withdrawn at screening were analyzed in the group to which they were originally assigned. Missing data from the mITT analysis was handled using multiple imputation via chained equations and included stratum, group assignment and baselines variable that met a minimum Kendall's tau of 0.2 with the primary outcome. No data was collected at 6 months 34 days for the Docudrama arm.
Measure: Count of Participants; unit: Participants
Groups:
- Docudrama: Participants were exposed to a docudrama related to blood donation.
Arm/Group | FRD: Control | VNRBD: Control | FRD:WhatsApp | VNRBD: WhatsApp | Docudrama
Number analyzed (Participants) | 27 | 30 | 28 | 31 | 0
Participants | 2 | 2 | 2 | 7 | 0
Statistical Analysis 1: Comparison: FRD: Control vs VNRBD: Control vs FRD:WhatsApp vs VNRBD: WhatsApp; The primary analysis applies only to the RCT participants (N=130). Docudrama participants were not assessed for return blood donation. Analysis used fitted logistic regression with outcome donation attempted (Y/N) on the modiﬁed intention-to-treat (mITT) population, adjusted for type of donor (FRD, VNRBD); Test type: Superiority; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.61 to 8.50] — The estimated odds ratio of return donation attempt represents WhatsApp compared to control; Missing data on the primary outcome from the mITT analysis was handled using multiple imputation via chained equations with 50 imputations, and included stratum, group assignment (WhatsApp, Control) and ethnicity. Ethnicity was the only baseline variable with a minimum Kendall's tau of 0.2 with donation attempt

ADVERSE EVENTS:
Time Frame: Participants were followed for serious adverse events (SAEs) from randomization until completion of follow-up, for a total of 6 months and 34 days. No SAEs were reported.
Groups:
- FRD Control: FRD Control: Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
- VNRBD Control: VNRBD Control: Participants in this group will receive the standard NBSG communications for first-time donors: 1) a thank you phone call and 2) and a reminder phone call two-weeks prior to the second blood donation eligibility. The second blood donation eligibility is four months after the first donation.
Arm/Group | FRD Control | VNRBD Control | FRD WhatsApp | VNRBD WhatsApp | Docudrama
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30 | 0/28 | 0/31 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30 | 0/28 | 0/31 | 0/14
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30 | 0/28 | 0/31 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The C-CAD pilot study was part of the BLOODSAFE initiative. The Publications and Presentations (P&P) Committee reviews and approves all abstracts, presentations, and manuscripts that utilize data generated from BLOODSAFE. The BLOODSAFE P&P Committee has voting members from the sponsor (NHLBI), the data coordinating center and each of the country-specific research teams (Ghana, Kenya, Malawi).

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT04783077/Prot_SAP_ICF_000.pdf